CLINICAL TRIAL: NCT03702400
Title: Randomized Double-blinded Comparison of Norepinephrine and Phenylephrine in Bolus for Maintenance of Blood Pressure During Spinal Anesthesia for Cesarean Delivery
Brief Title: Norepinephrine or Phenylephrine in Bolus for Hypotension in Cesarean Delivery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital dos Servidores do Estado do Rio de Janeiro (Other Government)
Responsible Party: Principal Investigator, DANIEL VIEIRA DE QUEIROZ, Department Chair, Hospital dos Servidores do Estado do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 000.603
Record Dates: First submitted 2018-10-06; First posted 2018-10-11 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Hypotension; Spinal Anesthesia
Keywords: phenylephrine; norepinephrine; cesarean delivery under spinal anesthesia
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine; Norepinephrine

STUDY DESIGN:
Intervention Model Description: In a randomized, double-blinded study, 76 healthy patients having cesarean delivery under spinal anesthesia will be randomized, using an electronic system (the Randomizer App®, Version 3.2 Wisse Keizer program), to have systolic blood pressure maintained with bolus of phenylephrine at a dose of 100 mcg bolus (at a dilution containing 20 mcg / mL), or with norepinephrine at a dose of 5 mcg (at a dilution containing 1 mcg / mL).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Phenylephrine 100 mcg (Active Comparator): Phenylephrine will be used at a dose of 100 mcg bolus at a dilution containing 20 mcg / mL of the drug to be used whenever systolic blood pressure falls below 10% of baseline.
  Interventions: Drug: Phenylephrine 100 mcg
- Norepinephrine 5 mcg (Experimental): Norepinephrine will be used at a dose of 5 mcg at a dilution containing 1 mcg / mL to be used whenever systolic blood pressure falls below 10% of baseline.
  Interventions: Drug: Norepinephrine 5 mcg

INTERVENTIONS:
Drug: Phenylephrine 100 mcg — Phenylephrine at a dose of 100 mcg bolus at a dilution containing 20 mcg / mL of the drug, 5 mL each bolus
  Other Names: Fenilefrin
  Arms: Phenylephrine 100 mcg
Drug: Norepinephrine 5 mcg — Norepinephrine at a dose of 5 mcg at dilution containing 1 mcg / mL, 5 mL each bolus
  Other Names: Hemitartarato de norepinefrina
  Arms: Norepinephrine 5 mcg

SUMMARY:
This study evaluate the ability of phenylephrine and of noradrenaline to maintain normal systemic arterial blood pressure and heart rate in healthy pregnant women submitted to cesarean section with spinal anesthesia. Half of participants will receive bolus of phenylephrine while the other half will receive bolus of noradrenaline.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, comparative two-group clinical study to observe two vasopressor drugs, phenylephrine and noradrenaline, in the ability to maintain systemic arterial pressure in pregnant women after spinal anesthesia for cesarean section; based on the hypothesis that, since noradrenaline has a predominant alpha-adrenergic action and a weak 1- beta-adrenergic beta action, it could be as capable of maintaining blood pressure effectively as phenylephrine, but with a lower frequency of bradycardia; patients who meet the inclusion criteria will be randomly assigned to one of the groups to be studied: group F - phenylephrine at a dose of 100mcg bolus and N - noradrenaline at the dose of 5mcg. One of these drugs will be used whenever systolic blood pressure drops below 10% of the baseline, additional doses will be allowed whenever necessary, aiming at maintaining the systolic blood pressure at baseline values; the blood pressure will be measured non-invasively and the heart rate by pulse oximeter and electrocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, with single gestation, with cesarean programming to be performed under spinal anesthesia;
* Age above 18 years;
* Physical State American Society of Anesthesiologists (ASA) II and III;
* Weight between 50kg and 120kg;
* Height between 140cm and 180cm.

Exclusion Criteria:

* Refusal to participate in the study;
* Pregnant women with fetus with known abnormalities;
* Pregnant women with cardiovascular disease;
* Pregnant women with pregnancy-specific hypertensive disease;
* Allergy to any medication to be used in the study;
* Users of monoamine oxidase inhibitors;
* Users of tricyclic antidepressants;
* Emergency caesarean section due to acute fetal distress;
* Situations in which the sensory level after single intrathecal injection of the local anesthetic does not reach at least T6 within 5 minutes after spinal anesthesia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Number of bolus required | during the procedure
  Number of bolus doses of phenylephrine and noradrenaline to maintain systemic arterial pressure at 90% of baseline in pregnant women undergoing spinal anesthesia for cesarean
Heart rate | during the procedure
  Number of episodes of heart rate under 60 bpm while using phenylephrine and noradrenaline in pregnant women undergoing spinal anesthesia for cesarean

SECONDARY OUTCOMES:
Neonatal gasometric outcome | during the procedure
  To evaluate the neonatal outcome through the analysis of venous and arterial blood gases collected in the cord umbilical after birth.
Neonatal Apgar outcome | during the procedure
  To evaluate the neonatal outcome through the classification given by the neonatologist responsible for the care to the newborn in the delivery room with the use of the Apgar Scale (0-10), 10 the better classification.
Nausea and vomiting | during the procedure
  To evaluate the incidence of nausea and vomiting of the parturient during cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: DANIEL V DE QUEIROZ, Principal Investigator — HOSPITAL FEDERAL DOS SERVIDORES DO ESTADO
Locations (1):
- Hospital Federal Dos Servidores Do Estado, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ngan Kee WD, Lee SW, Ng FF, Tan PE, Khaw KS. Randomized double-blinded comparison of norepinephrine and phenylephrine for maintenance of blood pressure during spinal anesthesia for cesarean delivery. Anesthesiology. 2015 Apr;122(4):736-45. doi: 10.1097/ALN.0000000000000601. PMID 25635593
- [Background] Vallejo MC, Attaallah AF, Elzamzamy OM, Cifarelli DT, Phelps AL, Hobbs GR, Shapiro RE, Ranganathan P. An open-label randomized controlled clinical trial for comparison of continuous phenylephrine versus norepinephrine infusion in prevention of spinal hypotension during cesarean delivery. Int J Obstet Anesth. 2017 Feb;29:18-25. doi: 10.1016/j.ijoa.2016.08.005. Epub 2016 Aug 28. PMID 27720613